CLINICAL TRIAL: NCT00535041
Title: Pilot Trial of Pre-operative Chemo/RT Using Xeloda and External Beam RT Followed by Definite Surgery in Patients With Localized Rectal CA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC#2011-031
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2016-01

CONDITIONS: Rectal Neoplasms
Keywords: Pilot trial of pre-operative chemo/RT using Xeloda and external beam RT followed by definite surgery in patients with localized rectal CA
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Chemotherapy, radiation therapy & surgery — radiation and chemotherapy

SUMMARY:
Pilot trial of pre-operative chemo/RT using Xeloda and external beam RT followed by definite surgery in patients with localized rectal CA

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized rectal CA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
safety | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shouki Bazarbashi, MD, Principal Investigator — KFSH&RC
Locations (1):
- KFSH&RC, Riyadh, Saudi Arabia